CLINICAL TRIAL: NCT04737733
Title: Effects of a Dementia-friendly Program on Detection and Management of Patients With Cognitive Impairment and Delirium in Acute-care Hospital Units: a Non-equivalent Control Group Design
Brief Title: Effects of a Dementia-friendly Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Nina Mickelson Weldingh, Prinsipal Investigator, University Hospital, Akershus
Organization: Oslo and Akershus University College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/666(REK)
Record Dates: First submitted 2021-01-26; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Delirium; Cognitive Impairment; Dementia
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: A non-equivalent control group design with a historical control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The dementia friendly hospital program (Other): The dementia-friendly hospital program comprised three parts; 1) Educational program for health practitioners to increase the staff's knowledge and awareness of patients with cognitive impairment and/or delirium; 2) Screening, for early identification of cognitive impairment and delirium, using the Four Assessment Test (4AT); 3) Delirium risk factor modification and management for patients defined with potential cognitive impairment and risk of delirium, implying that risk factor modifications should be implemented in the patient's care plan. For patients with suspected delirium, the program promoted an additional delirium management plan.
  Interventions: Other: The dementia friendly program

INTERVENTIONS:
Other: The dementia friendly program — Implementation of a systematic screening and risk modification and management plan, to identify and enhance the management of patients with cognitive impairment and risk of delirium.

SUMMARY:
Frail older persons with cognitive impairment are at special risk of experiencing delirium during acute hospitalisation. The purpose of this study was to investigate whether a dementia-friendly hospital program contributes to improved detection and management of patients with cognitive impairment and delirium.

DETAILED DESCRIPTION:
Study design This study, has a non-equivalent control group design and a historical control Group. The Control group received usual care and the experimental group received usual care plus the dementia-friendly program.

One Group received care after implementing the dementia-friendly hospital program. The study is performed at two medical wards at a large acute-care hospital in Norway. A medical pulmonary ward and a cardiac ward participated.

Data Collection:

Demographic data included age, gender, place of residence (home, adapted housing, institution), and family/relative network, and were obtained upon admission to the study.

Medical data included cause of admission, active medical diagnoses, medications and medical treatment, and were obtained both at admission and from their electronic medical records after discharge.

Cognitive Impairment and delirium were assessed with two different screening tools: the Four Assessment Test (4AT) and the Confusion Assessment Method (CAM).

For all patients with a positive 4AT (≥1) or identified cognitive impairment during their hospital stays, a thorough review of the patient's journal was conducted upon discharge to record if, in case of yes, which type of preventive or treatment measures according to the dementia-friendly program, the patients had received during their stays.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥75 years
* acute admission to the cardiac or pulmonary wards.
* Patient who has given informed written consent, or proxy consent from relatives for patients who lacked cognitive capacity.

Exclusion Criteria:

* Readmitted patients enrolled in a previous hospital stay.
* Patients who do not have sufficient verbal function or hearing to communicate
* Patients in a coma or too ill to participate
* Patients who are isolated
* Patients who do not wish to participate or relatives who do not want the patient to participate, in the cases where the patient lacked cognitive capacity to consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 423 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Detection of patients with cognitive impairment | During the stay at the participating wards, assessed from the electronical medical record within 6 months after discharge
  Proportion of patients identified with cognitive impairment during the hospital stay, documented in the electronic Medical record. Difference between the control group and the intervention group. Patients were assessed with The Four Assessment Test at admission and during the stay at the participating wards. Furthermore, documentation of cognitive impairment in the electronic medical journal during the stay were assessed after discharge.
Management of patients with cognitive impairment and delirium | During the stay at the participating wards, assessed from the electronical medical record within 6 months after discharge
  Proportion of patients identified with cognitive impairment, delirium or at risk of delirium who has documented interventions to prevent and/or treat delirium, according to the implemented dementia-friendly program.Differences between the control group and the intervention group.

SECONDARY OUTCOMES:
Screening within 24 hours | Within 24 hours after admission to the ward
  Proportion of patients screened with The Four Assessment Test within 24 after hours after admission to the ward. Differences between the control group and the intervention group.
Use of antipsychotics, hypnotics and sedatives | During the stay at the participating wards, assessed from the electronical medical record within 6 months after discharge
  Proportion of patients with cognitive impairment given doses of antipsychotics, hypnotics and sedatives during the stay at the participating wards. Differences between the control group and the intervention group. Given doses of antipsychotics, hypnotics and sedatives during the stay at the participating wards registered in the electronic medical journal, were assessed after discharge.
Use of medications not recommended for the patient group | During the stay at the participating wards, assessed from the electronical medical record within 6 months after discharge
  Proportion of patients with cognitive impairment who uses medications which are not recommended for the patient group. Differences between the control group and the intervention group.
Departure to rehabilitation or nursing home | Assessed from the electronical medical record, within 6 month after discharge
  Proportion of patients with departure to rehabilitation or nursing home. Departure to care level were assessed from the electronic medical journal after discharge.Differences between the control group and the intervention group.
Length of hospital stay | Assessed from the electronical medical record, within 6 month after discharge
  Mean number of days at the hospital stay.Length of hospital stay were collected from the electronic medical journal after discharge.Differences between the control group and the intervention group.
Delirium | Assessed from the electronical medical record, within 6 month after discharge
  Proportion of patients diagnosed with delirium. Delirium diagnosis documented during the stay at the participating wards were collected from the electronical medical record after discharge. Differences between the control group and the intervention group.
30-day readmission to the hospital | Readmissions to the hospital were assessed from the electronical medical record 30 days after discharge.
  Proportion of patients who are readmitted to the hospital within 30 days after discharge from the hospital. Differences between the control group and the intervention group.
30-day mortality | Mortality were assessed from the electronical medical record 30 days after discharge.
  Proportion of mortality in the patient group within 30 days after discharge from the hospital. Differences between the control group and the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Nina M Weldingh, Master, Principal Investigator — University Hospital, Akershus
Locations (1):
- University hospital, Akershus, Lørenskog, Norway

REFERENCES:
- [Derived] Weldingh NM, Mellingsaeter MR, Hegna BW, Benth JS, Einvik G, Juliebo V, Thommessen B, Kirkevold M. Impact of a dementia-friendly program on detection and management of patients with cognitive impairment and delirium in acute-care hospital units: a controlled clinical trial design. BMC Geriatr. 2022 Mar 31;22(1):266. doi: 10.1186/s12877-022-02949-0. PMID 35361136